CLINICAL TRIAL: NCT01982318
Title: A Prospective, Multi-Center, Randomized, Double Blind, Placebo-Controlled Trial Comparing Vitrogro® ECM To Placebo As An Adjunct To Standard Care In Patients With Venous Leg Ulcers
Brief Title: A Prospective Randomized, Double-Blind, Placebo-Controlled Trial Comparing VitroGro® ECM to Placebo in Patients With Venous Leg Ulcers
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study discontinued. Superseded by NCT02973893 VF00102.
Sponsor: Tissue Therapies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vitro-US-1001
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Venous Leg Ulcer
Keywords: Venous Leg Ulcer; Leg Ulcer; Venous Hypertension; Venous Reflux; Deep Venous System; Chronic leg ulceration; Calf perforator
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VitroGro®ECM (Active Comparator): A topical application of synthetic extracellular matrix (ECM) protein formulation to the wound bed) plus Standard Care (moisture retentive dressing and multi-layer compression therapy).
  Interventions: Drug: VitroGro® ECM
- Dulbecco's Phosphate Buffered Saline (Placebo Comparator): Dulbecco's Phosphate Buffered Saline plus Standard Care (moisture retentive dressing and multi-layer compression therapy).
  Interventions: Drug: Dulbecco's Phosphate Buffered Saline

INTERVENTIONS:
Drug: VitroGro® ECM
  Arms: VitroGro®ECM
Drug: Dulbecco's Phosphate Buffered Saline
  Arms: Dulbecco's Phosphate Buffered Saline

SUMMARY:
The objective of this study is to assess the efficacy and safety of VitroGro® combined with standard care in the treatment of Venous Leg Ulcers (VLUs) compared to Placebo with standard care over the course of the 8-week treatment phase.

ELIGIBILITY:
Abbreviations:

* Study Ulcer: SU
* Post-debridement: PD

Inclusion Criteria: Potential subjects are required to meet all of the following criteria for enrollment into the study and subsequent randomization.

1. 18≤ years old.
2. Ankle Brachial Pressure Index ≥0.80. (Calculations made using measurements from posterior tibial & dorsalis pedis arteries & both arms).
3. Presence of a venous leg ulcer extending through the full thickness of the skin, but not down to muscle, tendon, or bone. The largest ulcer will be designated the SU and the only one included in the study. If other ulcerations are present on the same leg they must be more than 2 cm apart from the SU.
4. Venous disease confirmed by Doppler ultrasound to demonstrate reflux of > 0.5 seconds in saphenous (great or small), calf perforators or the deep venous system. Subjects with prior venous surgery may be included if they still demonstrate significant reflux in a remaining venous segment and the SU continues to suffer poor healing because of venous hypertension.
5. SU has been present 1 ≤ x ≤ 12 months prior to the initial screening visit, and is excluded if it has undergone 12 months of continuous high strength compression therapy over its duration.
6. SU with a 2.5 ≤ x ≤ 20 cm2 at the T1 visit (PD).
7. SU with a clean, granulating base free of adherent slough at the T1 visit (PD).
8. In the case of a female patient of childbearing potential, willingness to use acceptable methods of contraception. A urine pregnancy test at the T1 visit must be administered, and must be negative for inclusion.
9. Understanding of and willingness by the patient to participate in the clinical study and ability to comply with study procedures and study visit schedule.
10. Reading, approval, and signature by the patient of the IRB/IEC ICF before screening procedures are undertaken.

Exclusion Criteria:Potential subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomization:

1. Ulcer(s) deemed by the Investigator to be caused by a medical condition other than venous insufficiency. These may include, but are not limited to: ulcerations due to fungal, malignant, diabetic, and/or arterial insufficiency causes.
2. Ulcer exhibits clinical signs and symptoms of infection at S1 or T1. The infection should be treated & afterward the patient may be re-assessed for eligibility for study re-entry.
3. Known allergy to any of the protocol-stipulated treatment procedures or non-tolerance of multi-layer compression therapy.
4. Ulcer, in the opinion of the Investigator, is suspicious for cancer.
5. A history of more than 2 weeks treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1 month prior to S1, or treatments with such medications during screening, or anticipated requirement of such medications during the course of the study.
6. Treatment with any investigational drug(s) or therapeutic device(s) within 30 days preceding S1; or anticipated use of any of these therapies during the course of the study.
7. Malignant disease not in remission for 5 or more years, other than basal cell or squamous cell carcinomas of the skin that have been medically or surgically treated without evidence of metastases.
8. History of radiation at the SU site.
9. As determined by medical history, presence of one or more medical conditions including renal, hepatic, hematologic, active auto-immune or immune diseases that, in the opinion of the Investigator, would make the subject an inappropriate candidate for this ulcer healing study.
10. Known history of having AIDS or history of HIV infection.
11. Previous participation in any VitroGro® ECM trial within the past 6 months.
12. SU has been previously treated with tissue engineered materials or other scaffold materials within 30 days prior to S1.
13. SU which in the opinion of the Investigator might require negative pressure wound therapy or hyperbaric oxygen during the course of the trial.
14. Presence of any condition(s) that seriously compromise(s) the subject's ability to complete this study, or a known history of poor adherence with medical treatment.
15. NYHA Class III and IV congestive heart failure (CHF), as defined by the following criteria:

    * Class III: Symptoms with moderate exertion
    * Class IV: Symptoms at rest
16. Uncontrolled Diabetes Mellitus, as measured by an HbA1c >10%.
17. Ulcer on the dorsum of the foot or with more than 50% of the ulcer below the malleolus is excluded.
18. Pregnancy or breast-feeding.
19. Increase or decrease by >30% in the SU surface area at the T1 visit (PD) as compared to the SU surface area as measured at the S1 visit (PD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound closure within Treatment Phase | 8 weeks
  The primary efficacy endpoint for the study is the time to complete wound closure, within the 8-week Treatment Phase, as assessed by the investigator. Complete wound closure is defined as 100% re-epithelialization with no presence of scab or drainage as assessed by the Investigator at PH0 and confirmed at PH2.
  The date of complete healing is defined as the date of the first assessment of complete closure (100% re-epithelialization with no presence of scab or drainage) when complete wound closure is confirmed at a study visit 14 days (±3 days) later. For the purposes of this study, the initial assessment of complete closure will occur at PH0 and complete closure will be confirmed at PH2.

SECONDARY OUTCOMES:
Percentage (%) change from baseline in ulcer surface area at the end of the Treatment Phase, as measured by SilhoutteStarTM | 8 weeks
Incidence of complete healing within Treatment Phase, as determined by Investigator assessment | 8 weeks
Incidence of complete healing at each visit within the 8-week Treatment Phase, as determined by Investigator assessment | 8 weeks
Percentage (%) surface area reduction from baseline, at each visit within the 8-week Treatment Phase, as measured by SilhoutteStarTM | 8 weeks
Time to first instance of no pain (i.e., pain score less than 5mm on VAS) | 12 weeks
Time to first instance when the patient expectation was met as assessed by Patient Benefit Index | 12 weeks
Incidence of ulcer recurrence, at the site of the ulcer, during the Post-Healing Phase | Up to 4 weeks post-treatment
Change in Quality of Life metrics at study end. | 12 weeks